CLINICAL TRIAL: NCT00015665
Title: Open-Label, Non-Comparative Protocol for the Emergency Use of Voriconazole in Patients With Life Threatening, Invasive Mycoses Who Are Failing on Currently Available Antifungal Agents
Brief Title: Emergency Use of Voriconazole in Patients With Life-Threatening Invasive Fungal Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010150; 01-I-0150
Record Dates: First submitted 2001-04-28; First posted 2001-04-30 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-03

CONDITIONS: Mycoses
Keywords: Fungal; Immunodeficiency; Infection; Refractory; Severe; Fungal Infections
MeSH Terms: conditions — Mycoses; Immunologic Deficiency Syndromes; Infections; Lymphoma, Follicular | interventions — Voriconazole

INTERVENTIONS:
Drug: Voriconazole

SUMMARY:
This protocol provides for emergency treatment with the experimental anti-fungal drug voriconazole for patients with life-threatening invasive fungal infections. The increase in the number of patients whose immune function is suppressed because of chemotherapy, tissue or organ transplantation, or HIV infection has led to an increase in fungal infections. New drugs are needed to combat these infections in patients who do not respond to or cannot tolerate standard treatments.

Patients on other primary NIH protocols who have an invasive life-threatening fungal infection that does not respond to currently available treatments or who cannot tolerate these treatments may be eligible for this study.

Participants will have a blood test and a physical examination before receiving voriconazole. They will receive voriconazole twice a day either as an infusion into a vein or as tablets taken by mouth. Adult patients will be asked to provide a blood sample any time after the first dose of voriconazole to be used for developing a test to measure voriconazole concentration in the blood. Patients will be evaluated about 10 days after starting treatment and then at least once every 4 weeks with a symptom check and blood test.

DETAILED DESCRIPTION:
The increase in the number of immunosuppressed patients as a result of more aggressive chemotherapy, transplantation, HIV infection has lead to an increase in the incidence of invasive fungal infections. Moreover, despite the availability of newer, less toxic preparations of Amphotericin B and azole antifungals such as fluconazole and itraconazole, invasive mycoses remain a therapeutic challenge.

Voriconazole is a new triazole that has shown in phase II studies to be very active against Aspergillus sp. Its side effect profile has been very benign, comparable with those of other FDA approved triazoles. In vitro studies also show that voriconazole has a very broad spectrum ranging from opportunistic to endemic fungi. In addition, the availability of intravenous and oral formulations add to its potential advantages because the therapy of these infections usually require long courses on antifungals.

In this study, voriconazole is used as a salvage therapy for those patients who are unable to tolerate or who have failed other antifungal therapies. Because of the abundance of immunocompromised patients at our center, we believe that having such a protocol ready for enrollment would mitigate delays in such crucial moments. We seek to enroll and treat 40 patients over a 3 year period.

ELIGIBILITY:
INCLUSION CRITERIA:

All subjects must have a proven fungal infection that is resistant to standard therapy, or to which the patient is significantly intolerant. (Intolerance must include signs of intolerance such as fever, rigors, laboratory abnormalities, as well as subjective symptoms).

Children are eligible.

EXCLUSION CRITERIA:

AST, ALT greater than 10x the upper limit of normal

Previous hypersensitivity to azole antifungals

Concomitant Rifampin, carbamazepine, or barbiturates or greater than 3 days of such drugs in the 14 days prior to treatment with voriconazole

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2001-04; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States